CLINICAL TRIAL: NCT00127439
Title: Differential Effects of Robotic vs. Manually-Assisted Locomotor Training
Brief Title: Effects of Robotic Versus Manually-Assisted Locomotor Training for Individuals With Incomplete Spinal Cord Injury
Acronym: DE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B4024-I
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Spinal Cord Injuries
Keywords: Ambulatory Disability; Disability Ambulation; Locomotion Disorders; Motor Activity; Rehabilitation; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robotic Assisted Locomotor Training (Experimental): A robotic stepping device in concert with a body weight support system and treadmill is used by a physical therapist and trainers for the participant with spinal cord injury to intensely practice task-specific standing and stepping to advance retraining the capacity to step. The robotic device provides the appropriate kinematics associated with standing and stepping.
  Interventions: Other: Robotic Assisted Locomotor Training
- Manually Assisted Locomotor Training (Experimental): A body weight support system and treadmill is used by a physical therapist and trainers for the participant with spinal cord injury to intensely practice task-specific standing and stepping to advance retraining the capacity to step. Therapists and trainers promote the appropriate kinematics associated with standing and stepping.
  Interventions: Procedure: Manually Assisted Locomotor Training

INTERVENTIONS:
Procedure: Manually Assisted Locomotor Training — The total program is 45 sessions, 5x/week with total locomotor training (LT) duration of 30 stepping minutes/day. 1) BWS is initiated at 40% and gradually decreasing to 0%, 2) treadmill speed is set at normal walking speeds and increased as tolerated, and 3) manual assistance given when the subject is unable to independently step or control upright posture, and decreased as participant progresses. Trainers assist via verbal cues and manual assistance to achieve good stepping. The goal for endurance is 20 mins of continuous, independent, coordinated stepping on the treadmill at 0% BWS. Participants are encouraged to assist and/or independently maintain an upright posture, weight shift onto the loaded limb, flex or extend their legs, and to swing their arms in coordination with the legs.
  Other Names: manually assisted body-weight supported treadmill training
  Arms: Manually Assisted Locomotor Training
Other: Robotic Assisted Locomotor Training — The total program is 45 sessions, 5x/week with total locomotor training (LT) duration of 30 stepping minutes/day. 1) BWS is initiated at 40% and gradually decreasing to 0%, 2) treadmill speed is set at normal walking speeds and increased as tolerated, and 3) manual assistance given when the subject is unable to independently step or control upright posture, and decreased as participant progresses. Trainers assist via verbal cues and manual assistance to achieve good stepping. The goal for endurance is 20 mins of continuous, independent, coordinated stepping on the treadmill at 0% BWS. Participants are encouraged to assist and/or independently maintain an upright posture, weight shift onto the loaded limb, flex or extend their legs, and to swing their arms in coordination with the legs.
  Other Names: robotic assisted body-weight supported treadmill training
  Arms: Robotic Assisted Locomotor Training

SUMMARY:
The purpose of this study is to collect data comparing two means of providing locomotor training: manual and robotic and the possible differential effects it may have on walking ability for persons with spinal cord injury (SCI).

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is one of the most disabling health problems facing adults today, with one of the consequences often being inability to walk or difficulty walking. Recent studies suggest that intensive step training on a treadmill using body-weight support (BWS) and manual assistance that provides repetitive task-specific sensory cues to the neural axis can improve the recovery of walking for persons with incomplete SCI. More recently, robotics have been developed as an alternative to manually-assisted training. Robotic-assisted training may allow for increased intensity of training, improve the reproducibility and consistency of training, and reduce the personnel needed to implement the training. However, the effects of robotic-assisted training compared to manually-assisted training are not known. An improved understanding of these differential effects and the mechanisms of improvement in walking can facilitate continued advances in evidenced-based practice of neuro-rehabilitation, therefore improving the treatment of persons with SCI.

The primary objective of this project is to assess and compare the effects of robotic-assisted versus manually-assisted locomotor training (LT) using the body-weight support (BWS) on sub-tasks of walking. Specifically, we believe that at least four sub-tasks of walking are differentially affected by the robotic-assisted training when compared to manually-assisted training (propulsion, transition from stance to step, stepping, and equilibrium). The investigators hypothesize that robotic-assisted training will have a greater effect on improving propulsion, transition and equilibrium. The effect of these two modalities on adaptability, a fifth sub-task of walking, is unclear; therefore, a development component of the pilot project will involve establishing a quantitative measure of adaptability and assessing differential effects of training. Participants will be randomized to one of two training groups: robotic-assisted or manually-assisted, and evaluated for performance on sub-tasks of walking.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Spinal cord injury (SCO) at least 6 months since injury
* Motor I-SCI, upper motor neuron lesion only at cervical or thoracic levels
* A diagnosis of first time SCI including etiology from trauma, vascular, or orthopedic pathology
* SCI as defined by the American ASIA Impairment Scale categories C or D
* Medically stable condition that is asymptomatic for bladder infection, decubiti, osteoporosis, cardiopulmonary disease, pain, contractures or other significant medical complications that would prohibit or interfere with testing of walking function and training or alter compliance with the training protocol
* Documented medical approval from the participant's personal physician verifying the participant's medical status at time of enrollment
* Ability to walk a minimum of 30 feet with or without an assistive device, independently or with minimal assistance
* Over ground gait speed < 0.8 m/s
* Persons using anti-spasticity medication must maintain stable medication dosage during the study
* Able to give informed consent

Exclusion Criteria:

* Current participation in a rehabilitation program/research protocol that could interfere or influence the outcome measures of the current study
* History of congenital SCI (e.g. myelomeningocele, intraspinal neoplasm, Friedreich's ataxia) or other degenerative spinal disorders (e.g. spinocerebellar degeneration, syringomyelia) that may complicate the protocol
* Inappropriate or unsafe fit of the harness or robotic trainer due to the participant's body size and/or joint contractures or severe spasticity that would prohibit the safe provision of either training modality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Behrman, PT PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Behrman AL, Harkema SJ. Locomotor training after human spinal cord injury: a series of case studies. Phys Ther. 2000 Jul;80(7):688-700. PMID 10869131
- [Background] Barbeau H, Norman K, Fung J, Visintin M, Ladouceur M. Does neurorehabilitation play a role in the recovery of walking in neurological populations? Ann N Y Acad Sci. 1998 Nov 16;860:377-92. doi: 10.1111/j.1749-6632.1998.tb09063.x. PMID 9928326
- [Background] Hesse S, Uhlenbrock D. A mechanized gait trainer for restoration of gait. J Rehabil Res Dev. 2000 Nov-Dec;37(6):701-8. PMID 11321006
- [Background] Colombo G, Joerg M, Schreier R, Dietz V. Treadmill training of paraplegic patients using a robotic orthosis. J Rehabil Res Dev. 2000 Nov-Dec;37(6):693-700. PMID 11321005
- [Background] Hornby TG, Zemon DH, Campbell D. Robotic-assisted, body-weight-supported treadmill training in individuals following motor incomplete spinal cord injury. Phys Ther. 2005 Jan;85(1):52-66. PMID 15623362
- [Background] Trimble MH, Behrman AL, Flynn SM, Thigpen MT, Thompson FJ. Acute effects of locomotor training on overground walking speed and H-reflex modulation in individuals with incomplete spinal cord injury. J Spinal Cord Med. 2001 Summer;24(2):74-80. doi: 10.1080/10790268.2001.11753558. PMID 11587422
- [Result] Day KV, Kautz SA, Wu SS, Suter SP, Behrman AL. Foot placement variability as a walking balance mechanism post-spinal cord injury. Clin Biomech (Bristol). 2012 Feb;27(2):145-50. doi: 10.1016/j.clinbiomech.2011.09.001. Epub 2011 Oct 14. PMID 22000699
- See also: Click here for more information about this study: Differential Effects of Robotic vs. Manually-Assisted Locomotor Training — http://www.brrc.research.va.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred through James A. Haley Veterans' Hospital, Tampa, VA; North Florida/South Georgia Veterans Health System, Gainesville, FL; Paralyzed Veterans of America - Central Florida Chapter; Brooks Rehabilitation Hospital, Jacksonville, FL; Shands Rehab Hospital, Gainesville, FL; and the FL Brain and SCI Network.
Pre-assignment Details: No significant events relative to enrollment.
Period: Overall Study
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 19 subjects were enrolled; 2 subjects (1:Manual; 1: Robotic) did not complete as intervening medical issues would not permit them to meet the study protocol's requirement for training intensity; and 2 subjects' (Manual) data was insufficient for data analysis and thus eliminated from analysis.
Groups:
- Robotic Assisted Locomotor Training: Robotic Assisted Locomotor Training - The total program was 45 sessions, 5x/week with total a locomotor training duration minimum of 30 stepping minutes/day.This occurred using a robotic device to provide assistance for stepping and standing kinematics with partial body weight support on a treadmill.
- Manually Assisted Locomotor Training: Manually Assisted Locomotor Training: The total program was 45 sessions, 5x/week with total a locomotor training duration minimum of 30 stepping minutes/day.This occurred on a treadmill with partial body weight support and manual assist from 3-4 trainers to produce stepping and standing kinematics.
- Total: Total of all reporting groups
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.75 (10.01) | 37.57 (16.48) | 41.93 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
Chronicity (months) [Mean (Standard Deviation); unit: months] — Chronicity = number of months since injury.
  months | 18.81 (15.97) | 23.21 (24.84) | 20.87 (19.92)
Lower Extremity Motor Score (X/50) [Mean (Standard Deviation); unit: units on a scale] — : Lower Extremity Motor Score = Strength based on bilateral leg muscle strength across 5 muscle groups: hip flexors, knee extensors, ankle dorsiflexors, long toe extensors, and ankle plantar flexors and scored 0-5 for each muscle group. 0 is the lowest score and 5 is the highest score. 0=total paralysis and 5= active movement, against gravity and normal resistance. Twenty-five (25) is the highest score possible for each lower extremity and thus 50 is the highest score for bilateral limbs.
  units on a scale | 40 (9) | 37 (13) | 38 (10)
Walking of SCI II (x/20) [Mean (Standard Deviation); unit: units on a scale] — Walking Index for SCI II - lowest score = 0 and highest score is 20. 0 is does not walk with equipment, bracing or assist and 20 is walks without a brace or device or physical assist for 10 meters.
  units on a scale | 12 (4.41) | 12 (4.84) | 12 (4.41)
Overground walking self-selected velocity [Mean (Standard Deviation); unit: meters/sec] — Overground walking Self-selected walking speed is provided in meters/sec with usual adult walking speed at 1.2 m/sec.
  meters/sec | 0.35 (0.21) | 0.31 (0.27) | 0.34 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Self Selected Velocity on Treadmill
Description: Subjects walk on a treadmill with overhead safety mounted to laboratory ceiling while wearing a harness. Treadmill speeds adjusted to lower than overground walking speeds and adjusted to patient reaches a comfortable speed.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Robotic Assisted Locomotor Training: Robotic Assisted Locomotor Training - Individuals with chronic SCI, upper motor neuron lesions at cervical and thoracic levels, and able to walk 30 feet and over 0.8 m/sec walking velocity.
- Manually Assisted Locomotor Training: Manually Assisted Locomotor Training - Individuals with chronic SCI, upper motor neuron lesions at cervical and thoracic levels, and able to walk 30 feet and over 0.8 m/sec walking velocity.
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
m/s
  Baseline Treadmill Walking Speed | 0.24 (0.12) | 0.22 (0.15)
  Post-Intervention walking speed | 0.4 (0.18) | 0.39 (0.17)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — The power analysis indicated that when the mean difference equals to 1.2 times of standard deviation, a two-sided t-test at 0.05 level will have 80% power; and for a mean difference of 1.4 times of standard deviation the power increases to 91%. To test the null hypothesis that correlation will be 0 at 0.5 level, a two-sided test based on Fisher's Z transformation will yield a power of 89% in detecting correlations of 0.6 or above with n=24 or above; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Pearson correlation of gait speed changes with directional difference of standardized kinematic scores (i.e. foot trajectory toe-off - degrees, foot trajectory toe-off - % cycle, foot trajectory initial contact - degrees, foot trajectory range - degrees, propulsive impulse N-s, minimum thigh angle - flexion degrees, minimum hip angle - extension degrees, trunk angle mid-stance); Test type: Superiority or Other; p = 0.05, Wilcoxon rank sum test

2. Primary Outcome: Stepping: Foot Trajectory Toe-Off
Description: Foot angle in a global reference frame at the start of swing phase during treadmill walking at self-selected speed. The kinematic outcomes were first standardized as deviations from control subjects who walk at similar speed (i.e., deviation from the control mean divided by SD among control). Stepping was quantified by the change in orientation of the foot angle (in a global reference frame) from the beginning to the end of the swing phase (i.e., foot-off to foot-down). The values will be identified from the processed 3-D kinematics for each walking cycle and average across steps.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
degrees
  Baseline Standardized Toe Off | 2.58 (1.2) | 0.92 (2.68)
  Post-Intervention Standardized Toe Off | 3.56 (1.83) | -0.58 (2.11)
  Baseline Raw Foot Trajectory Toe Off | -23.17 (12.78) | -38.87 (24.98)
  Post LT Raw Foot Trajectory Toe-Off | -22.46 (11.44) | -53.52 (18.77)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.05, t-test, 2 sided

3. Primary Outcome: Stepping: Foot Trajectory Toe-off % Cycle
Description: The outcome measure is the percentage of the gait cycle (%) for the occurrence of toe off. Foot trajectory toe-off was identified as indicated in the prior primary outcome (#2). The occurrence of toe-off was then identified relative to the percent of a complete gait cycle and thus the end point of the stance component of the gait cycle and the point of initiation for the swing component of the gait cycle. This outcome is reported in per cent of gait cycle.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of gait cycle
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
percentage of gait cycle
  Standardized Baseline Foot Toe Off % Cycle | -0.46 (5.93) | 4.51 (3.35)
  Standardized Post-LT Toe off % cycle | -2.23 (4.88) | 1.02 (3.58)
  Raw Pre Toe Off % cycle | 74.1 (13.84) | 85.66 (8.06)
  Raw Post-LT Toe Off % cycle | 67.52 (11.36) | 75.38 (9.22)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Provided previously; p = 0.05, t-test, 2 sided

4. Primary Outcome: Foot Trajectory Initial Contact
Description: Foot trajectory initial contact is the foot angle in a global reference frame at the end of swing (start of stance phase) during treadmill walking at self-selected speed when the foot contacts the ground (i.e. heel strike, foot contact, initial contact). The kinematic outcomes were first standardized as deviations from control subjects who walk at similar speed (i.e. deviation from the control mean divided by the SD among control). Foot trajectory initial contact (heel strike) was quantified by the orientation of the foot angle (in a global reference frame) at foot down (initial contact or heel strike). The values will be identified from the process 3-D kinematics for each walking cycle and averaged across steps. The outcome measurement is in degrees.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
degrees
  Standardized Pre-LT Foot Initial Contact HS | -2.57 (1.55) | -3.94 (2.54)
  Post-LT Foot Initial Contact HS | -2.99 (3.15) | -4.23 (4.88)
  Raw Pre Foot Contact Initial HS | 0.71 (5.1) | -4.35 (9.62)
  Raw Post Foot Initial Contact HS | 0.5 (11.56) | -4.87 (18.96)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Provided previously; p = 0.05, t-test, 2 sided

5. Primary Outcome: Foot Trajectory Range (Toe Off to Heel Strike)
Description: Range of foot trajectory from toe off to heel strike in degrees. The kinematic outcomes were first standardized as deviations from control subjects who walk at similar speed (i.e., deviation from the control mean divided by SD among control).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
degrees
  Standardized Pre-LT Foot Trajectory Range | 2.14 (2.04) | -2.22 (5.06)
  Standardized Post-LT Foot Trajectory Range | 3.12 (3.22) | -2.98 (5.11)
  Raw Pre-LT Foot Trajectory | -10.06 (8.13) | -27.24 (19.62)
  Raw Post-LT Foot Trajectory | -9.41 (10.27) | -30.73 (19.3)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.05, t-test, 2 sided

6. Primary Outcome: Propulsion: Propulsive Impulse
Description: Push-off force at toe off in N-s during treadmill stepping
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: N-s
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
N-s
  Standardized Pre-LT Propulsive Force | 1.51 (2.77) | 7.76 (7.23)
  Standardized Post-LT Propulsive Force | 2.08 (4.37) | 7.12 (8.17)
  Raw Pre-LT Propulsive Force | 9.06 (3.75) | 15.97 (8.02)
  Raw Post-LT Propulsive Force | 8.48 (3.75) | 14.35 (9.48)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.05, t-test, 2 sided

7. Primary Outcome: Kinematics: Minimum Thigh Angle
Description: Greatest thigh angle for hip flexion during stepping
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Manually Assisted Locomotor Training: A body weight support system and treadmill is used by a physical therapist and trainers for the participant with spinal cord injury to intensely practice task-specific standing and stepping to advance retraining the capacity to step. Therapists and trainers promote the appropriate kinematics associated with standing and stepping.
  The goal for endurance is 20 mins of continuous, independent, coordinated stepping on the treadmill at 0% BWS. Participants are encouraged to assist and/or independently maintain an upright posture, weight shift onto the loaded limb, flex or extend their legs, and to swing their arms in coordination with the legs.
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
degrees
  Standardized Pre-LT Thigh Angle Flexion | 1.45 (2.58) | -0.33 (3.14)
  Standardized Post-LT Thigh Angle Flexion | 1.54 (2.84) | -1.71 (2.64)
  Raw Pre-LT Thigh Angle Flexion | -6.9 (8.24) | -12.4 (9.77)
  Raw Post-LT Thigh Angle Flexion | -7.23 (9.04) | -17.05 (8.22)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.05, t-test, 2 sided

8. Primary Outcome: Kinematics: Minimum Hip Angle - Extension
Description: Hip angle at maximal hip extension during stepping
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
degrees
  Standardized Pre-LT Minimum Hip Angle Extension | 0.11 (2.46) | -1.79 (2.27)
  Standarized Post-LT Min Hip Angle Extension | 0.74 (2.26) | -2.4 (2.31)
  Raw Pre-LT Min Hip Angle Extension | -0.09 (12.74) | -9.8 (11.54)
  Raw Post-LT Min Hip Angle Extension | 2.21 (12.32) | -13.78 (11.3)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.05, t-test, 2 sided

9. Primary Outcome: Kinematics: Trunk Angle Mid-Stance
Description: Trunk Angle Mid-Stance - position in degrees
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Number analyzed (Participants) | 8 | 7
degrees
  Standardized Pre-LT Trunk Angle Midstance | -1.41 (2.93) | -0.72 (2.86)
  Standardized Post-LT Trunk Angle Midstance | -1.84 (2.93) | -0.72 (2.86)
  Raw Pre-LT Trunk Angle Midstance | -10.79 (10.12) | -8.01 (12.01)
  Raw Post-LT Trunk Angle Mid-Stance | -9.73 (11.78) | -12.31 (12.02)
Statistical Analysis 1: Comparison: Robotic Assisted Locomotor Training vs Manually Assisted Locomotor Training; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 13 week total possible period for documentation of adverse events. During the 45 session period of daily locomotor training (5x/week for 9 consecutive weeks) and the one week of pre-testing and one week of post-testing, and up to two additional weeks of training if subject cancelled sessions for illness or otherwise.
Description: Systematic review of patient occurred for overall health/condition of skin, joints, health status at start and end of every session and throughout the training session.
Groups:
- Manually Assisted Locomotor Training: A body weight support system and treadmill is used by a physical therapist and trainers for the participant with spinal cord injury to intensely practice task-specific standing and stepping to advance retraining the capacity to step. The therapist and trainers manually provide the appropriate kinematics associated with standing and stepping.
Arm/Group | Robotic Assisted Locomotor Training | Manually Assisted Locomotor Training
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/10
Other Adverse Events (participants affected / at risk) | 6/9 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Assisted Locomotor Training (N=9) | Manually Assisted Locomotor Training (N=10)
Hospitalized (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Participant hospitalized with elevated temperature and elevated blood pressure. Diagnosed with sepsis in bloodstream; hospitalized over weekend, self-report.
Hospitalized (Infections and infestations) | 0 (0) | 1 (1) — Infected wound at base of sacrum.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Assisted Locomotor Training (N=9) | Manually Assisted Locomotor Training (N=10)
Dizzy (Vascular disorders) | 1 (1) | 1 (2) — Dizziness upon standing; circulatory
Skin abrasion (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (7) — Skin abrasion
Loss of balance/fall (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) — Loss of balance that took subject to the floor, no injury
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) — Knee and foot pain
Colored urine (Renal and urinary disorders) | 1 (2) | 1 (1) — Blood tinged urine
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
muscle pain groin (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle soreness (leg) (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (Infections and infestations) | 0 (0) | 1 (1)
Not feeling well (General disorders) | 0 (0) | 1 (1)
Pulled back muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Occurred over weekend; unrelated
Catheter loosens and comes off during training (General disorders) | 1 (1) | 0 (0) — Urine spillage due to incident.

LIMITATIONS AND CAVEATS:
Data for two subjects was incomplete during outcome measures acquisition, interpretable and removed from data analysis.Two subjects did not complete.

An n=24 was anticipated; an original N=19 enrolled, the group sizes decreased to 8 and 7.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No